CLINICAL TRIAL: NCT02121210
Title: An Open-label, Randomized, Parallel Group Study Assessing the Immunogenicity and Safety of Sarilumab Administered as Monotherapy in Patients With Active Rheumatoid Arthritis
Brief Title: To Evaluate the Immunogenicity and Safety of Sarilumab Administered as Monotherapy in Patients With Rheumatoid Arthritis (RA)
Acronym: SARIL-RA-ONE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Collaborators: Regeneron Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EFC13752; 2013-002790-22; U1111-1143-4344 (Other: UTN)
Record Dates: First submitted 2014-04-21; First posted 2014-04-23 (Estimated); Results first posted 2017-06-20 (Actual); Last update posted 2017-06-20 (Actual); Status verified 2017-05

CONDITIONS: Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — sarilumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sarilumab 150 mg q2w (Experimental): Sarilumab 150 mg subcutaneous (SC) injection every two weeks (q2w) for 24 weeks.
  Interventions: Drug: sarilumab SAR153191 (REGN88)
- Sarilumab 200 mg q2w (Experimental): Sarilumab 200 mg SC injection q2w for 24 weeks.
  Interventions: Drug: sarilumab SAR153191 (REGN88)

INTERVENTIONS:
Drug: sarilumab SAR153191 (REGN88) — Pharmaceutical form: Solution for injection; Route of administration: Subcutaneous

SUMMARY:
Primary Objective:

To evaluate the immunogenicity of sarilumab administered as monotherapy.

Secondary Objectives:

* To evaluate the other safety aspects of sarilumab administered as monotherapy.
* To assess the exposure of sarilumab administered as monotherapy.

DETAILED DESCRIPTION:
Total study duration was up to 34 weeks: Up to 4-week screening period, 24-week open-label treatment phase, 6-week post-treatment observation. After completion of the treatment phase of this study, participants were eligible to enter a long term safety study (LTS11210 - SARIL-RA-EXTEND) for continuous treatment with sarilumab (SAR153191 [REGN88]).

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of rheumatoid arthritis (RA) ≥ 3 months.
* Moderately to severely active rheumatoid arthritis.
* Participants who per investigator judgment were incomplete responders to at least 12 weeks of an adequate dose of continuous treatment with or who were intolerant of one or a combination of non-biologic disease modifying anti-rheumatic drugs (DMARDs).

Exclusion criteria:

* Participants < 18 years of age.
* Past history of, or current, autoimmune or inflammatory systemic or localized joint disease(s) other than RA.
* History of juvenile idiopathic arthritis or arthritis onset prior to age 16.
* Severe active systemic RA, including but not limited to vasculitis, pulmonary fibrosis, and/or Felty's syndrome.
* Prior treatment with any biologic anti-interleukin 6 (IL-6) or IL-6 receptor (IL-6R) antagonist therapies.
* Treatment with prednisone > 10 mg or equivalent per day, or change in dosage within 4 weeks prior to randomization.
* New treatment with or dose-adjustment of on-going nonsteroidal anti-inflammatory drug (NSAIDs) or cyclooxygenase-2 (COX-2) inhibitors within 4 weeks prior to randomization, except for the use of low-dose acetylsalicylic acid for cardiovascular diseases.
* Use of parenteral glucocorticoids or intra-articular glucocorticoids injection within 4 weeks prior to randomization.
* Prior treatment with a Janus kinase (JAK) inhibitor (tofacitinib).
* New treatment or dose-adjustment to on-going medication for dyslipidemia, such as statin, within 6 weeks prior to randomization.
* Participation in any clinical research study evaluating another investigational drug or therapy within 5 half-lives or 60 days of first dose of study drug administration, whichever is longer.
* Participants with a history of malignancy other than adequately-treated carcinoma in-situ of the cervix, non-metastatic squamous cell or basal cell carcinoma of the skin, within 5 years prior to the randomization visit. Non-malignant lymphoproliferative disorders are also excluded.
* Participants with active tuberculosis or untreated latent tuberculosis infection.
* Pregnant or breast feeding women.

The above information is not intended to contain all considerations relevant to a Participant's potential participation in a clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Actual)
Dates: Start 2014-06; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (28):
- United States (13):
  - Investigational Site Number 840072, Gilbert, Arizona
  - Investigational Site Number 840049, Upland, California
  - Investigational Site Number 840220, South Miami, Florida
  - Investigational Site Number 840230, Elizabethtown, Kentucky
  - Investigational Site Number 840233, Minot, North Dakota
  - Investigational Site Number 840127, Oklahoma City, Oklahoma
  - Investigational Site Number 840011, Tulsa, Oklahoma
  - Investigational Site Number 840009, Duncansville, Pennsylvania
  - Investigational Site Number 840025, Jackson, Tennessee
  - Investigational Site Number 840032, Amarillo, Texas
  - Investigational Site Number 840074, Mesquite, Texas
  - Investigational Site Number 840124, Clarksburg, West Virginia
  - Investigational Site Number 840231, Franklin, Wisconsin
- Investigational Site Number 152002, Santiago, Chile
- Czechia (3):
  - Investigational Site Number 203034, Pardubice
  - Investigational Site Number 203001, Prague
  - Investigational Site Number 203002, Uherské Hradiště
- Estonia (2):
  - Investigational Site Number 233010, Tallinn
  - Investigational Site Number 233002, Tallinn
- Hungary (3):
  - Investigational Site Number 348014, Budapest
  - Investigational Site Number 348025, Budapest
  - Investigational Site Number 348021, Esztergom
- Poland (3):
  - Investigational Site Number 616018, Poznan
  - Investigational Site Number 616031, Warsaw
  - Investigational Site Number 616012, Wroclaw
- Russia (3):
  - Investigational Site Number 643006, Kemerovo
  - Investigational Site Number 643001, Moscow
  - Investigational Site Number 643016, Ryazan

REFERENCES:
- [Derived] Wells AF, Parrino J, Mangan EK, Paccaly A, Lin Y, Xu C, Fan C, Graham NMH, van Hoogstraten H, Torri A. Immunogenicity of Sarilumab Monotherapy in Patients with Rheumatoid Arthritis Who Were Inadequate Responders or Intolerant to Disease-Modifying Antirheumatic Drugs. Rheumatol Ther. 2019 Sep;6(3):339-352. doi: 10.1007/s40744-019-0157-3. Epub 2019 May 14. PMID 31090044

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 27 centers in 7 countries. A total of 201 participants were screened between 03 June 2014 and 20 October 2014.
Pre-assignment Details: Of 201 participants, 69 participants were screen failures due to exclusion criteria met and inclusion criteria not met. 132 participants were randomized in 1:1 ratio to either sarilumab 150 mg every two weeks (q2w) or sarilumab 200 mg q2w.
Groups:
- Sarilumab 150 mg q2w: Sarilumab 150 mg subcutaneous (SC) injection q2w for 24 weeks
Period: Overall Study
Arm/Group | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Started | 65 | 67
Completed | 58 | 58
Not Completed | 7 | 9
Not completed — Adverse Event | 5 | 7
Not completed — Lack of Efficacy | 2 | 0
Not completed — Other than specified above | 0 | 2

BASELINE CHARACTERISTICS:
Population: Randomized population that included any participant who signed an informed consent and was allocated to a randomized treatment regardless of whether the treatment kit was used or not.
Groups:
- Sarilumab 150 mg q2w: Sarilumab 150 mg SC injection q2w for 24 weeks.
- Total: Total of all reporting groups
Arm/Group | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w | Total
Number analyzed (Participants) | 65 | 67 | 132
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.1 (12.7) | 53.6 (14.1) | 52.4 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 57 | 106
  Male | 16 | 10 | 26

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Incidence of Antidrug Antibodies (ADA)
Description: ADA to sarilumab and anti-sarilumab neutralizing antibodies in serum samples were determined using a validated electrochemiluminescence immunoassay method. Percentage of participants with positive ADA during treatment emergent adverse event (TEAE) period (time from first dose of investigational medicinal product [IMP] to last dose of IMP + 60 days) was determined. Persistent ADA Response: treatment-emergent ADA detected at 2 or more consecutive sampling time points during the TEAE period, where the first and last ADA positive samples were separated by a period of at least 16 weeks or if the last measured sample was positive. ADA samples were collected prior to IMP administration at Week 0 (baseline), Week 2, 4, 12, 24 and 30.
Time Frame: From Baseline to Week 30 [End of study (EOS)]
Population: Analysis was performed on immunogenicity population included all randomized participants who received at least one dose of sarilumab with at least one post-dose, evaluable ADA sample.
Measure: Number; unit: Percentage of participants
Arm/Group | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 65 | 66
Percentage of participants
  Overall positive | 24.6 | 18.2
  Persistent positive | 12.3 | 6.1
  Persistent neutralizing positive | 10.8 | 3.0

2. Secondary Outcome: Serum Sarilumab Concentration
Description: Trough Concentration (Ctrough).
Time Frame: Pre-dose at Week 0 (Baseline), 2, 4, 12, 16, 20, 24 and 30
Population: Analysis was performed on pharmacokinetic (PK) population consisted of all randomized population actually received at least one or partial dose of IMP, with at least one post-dose, non-missing serum sarilumab concentration. Number of participants analyzed=participants with serum sarilumab concentration assessment at specified time-points.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sarilumab 150 mg q2w | Sarilumab 200 mg q2w
Number analyzed (Participants) | 54 | 52
ng/mL | 7350 (8030) | 17200 (15900)

ADVERSE EVENTS:
Time Frame: All adverse events (AEs) were collected from signature of the informed consent form up to the final visit (Week 30) regardless of seriousness or relationship to investigational product.
Description: Reported adverse events are treatment-emergent adverse events that is AEs that developed/worsened during the time from the first dose of IMP to last dose of IMP + 60 days.
Groups:
- Sarilumab 150mg q2w: Sarilumab 150 mg SC injection q2w for 24 weeks.
- Sarilumab 200mg q2w: Sarilumab 200 mg SC injection q2w for 24 weeks.
Arm/Group | Sarilumab 150mg q2w | Sarilumab 200mg q2w
Serious Adverse Events (participants affected / at risk) | 1/65 | 2/67
Other Adverse Events (participants affected / at risk) | 16/65 | 23/67
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sarilumab 150mg q2w (N=65) | Sarilumab 200mg q2w (N=67)
Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sarilumab 150mg q2w (N=65) | Sarilumab 200mg q2w (N=67)
Upper respiratory tract infection (Infections and infestations) | 3 | 4
Urinary tract infection (Infections and infestations) | 2 | 4
Neutropenia (Blood and lymphatic system disorders) | 8 | 11
Hypertension (Vascular disorders) | 0 | 4
Injection site erythema (General disorders) | 5 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If no publication has occurred within 12 months of the completion of the study, the Investigator shall have the right to publish/present independently the results of the study. The Investigator shall provide the Sponsor with a copy of any such presentation/publication for comment at least 30 days before any presentation/submission for publication. If requested by the Sponsor, any presentation/submission shall be delayed up to 90 days, to allow the Sponsor to preserve its proprietary rights.